CLINICAL TRIAL: NCT06687434
Title: Carb Counting vs. Simplified Qualitative Meal-Size Estimation- A Randomized Control Trial
Brief Title: Carb Counting vs. Simplified Qualitative Meal-Size Estimation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RMC-0411-24ctil
Record Dates: First submitted 2024-10-21; First posted 2024-11-13 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Automated insulin delivery system; carb counting
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accurate carb counting (Experimental): Participants will use precise carb counting to manage their meals
  Interventions: Behavioral: accurate carb counting
- Simplified qualitative meal-size estimation (Experimental): Participants will use a simplified meal announcement based on three presets for each meal, small, medium, or large, which will be personalized based on the dietitian assessment.
  Interventions: Behavioral: Simplified qualitative meal size estimation

INTERVENTIONS:
Behavioral: accurate carb counting — Participants will use precise carb counting to manage their meals
  Arms: Accurate carb counting
Behavioral: Simplified qualitative meal size estimation — participants will use a simplified meal announcement based on three presets for each meal, small, medium, or large, which will be personalized based on the dietitian's assessment.
  Arms: Simplified qualitative meal-size estimation

SUMMARY:
The goal of this study is to compare qualitative meal-size estimation to accurate carb counting in adolescents with Type One Diabetes using all available AID (Automated Insulin Delivery) systems. We will compare glucose control parameters and patient related outcome measures between the groups. 120 children and adolescents with type 1 Diabetes who begin using AID system will be randomly assigned to one of two groups: simplified qualitative meal size estimation or accurate carb counting. The study will last 6 months, with an additional optional follow up points at 12 and 24 months.

In the first visit all patients will receive nutrition guidance from the dietitian. In the accurate carb counting group, participants will use precise carb counting to manage their meals. In the simplified qualitative meal-size estimation group, participants will use a simplified meal announcement based on three presets for each meal, small, medium, or large, which will be personalized based on the dietitian's assessment. During the study, the dietitian will evaluate the insulin-to-carb ratio and meal estimation at least once in the first two weeks.

Follow-up visits will be scheduled at 4-6 weeks, 3, and 6 months after the study's initiation. At each visit participants will upload their data from their AID systems. Evaluation of their diabetes control will be made and an assessment regarding the carbohydrates calculation method. Digital questionnaires assessing diabetes distress, disordered eating behaviors, dietary regimen, and eating patterns will be provided at the beginning of the study and after 6 months, with an additional optional follow-up points that will be held at 12 and 24 months after the study's initiation.

ELIGIBILITY:
Inclusion Criteria:

1. T1D- diagnosed
2. Age 6-18 years
3. Treated with insulin (multiple daily injections or pump) and intending to initiate treatment with AID systems

Exclusion Criteria:

1. Non-T1D
2. Unstable medical conditions (other than diabetes) that may impact weight or diabetes management (as severe psychiatric disorders, various syndromes)
3. Use of medications that may impact weight or diabetes management (as use of steroids for an extended period of time. use of GLP-1)
4. Inability to understand the information, material and questionnaires of the study -

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in target range (70-18mg/dl) | Screening, after 4-6 weeks, after 3 months and after 6 months
Hemoglobin A1C | Screening, after 4-6 weeks, after 3 months and after 6 months
Percentage Continuous glucose monitoting usage | Screening, after 4-6 weeks, after 3 months and after 6 months
Number of Episodes of severe hypoglycemia | Screening, after 4-6 weeks, after 3 months and after 6 months
Number of episodes of Diabetic Ketoacidosis | Screening, after 4-6 weeks, after 3 months and after 6 months

SECONDARY OUTCOMES:
Total daily insulin dose | at screening, after 4-6 weeks, after 3 months and after 6 months.
basal insulin dose | at screening, after 4-6 weeks, after 3 months and after 6 months.
Number of manual boluses per day | at screening, after 4-6 weeks, after 3 months and after 6 months.
Number of announced meals per day | at screening, after 4-6 weeks, after 3 months and after 6 months.
Daily carbohydrates input | at screening, after 4-6 weeks, after 3 months and after 6 months.
Percentage of automated insulin delivery use | at screening, after 4-6 weeks, after 3 months and after 6 months.
Number of automated insulin delivery exits per week | at screening, after 4-6 weeks, after 3 months and after 6 months.
Percentage of automated boluses | at screening, after 4-6 weeks, after 3 months and after 6 months.
Score of Diabetes distress according to questionnaire | At screening and after 6 months
Score of Disordered eating behaviors according to quesiotnnaire | At screening and after 6 months
Score of Dietary regimen according to questionnaire | At screening and after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided